CLINICAL TRIAL: NCT00430443
Title: Phase I Study of Liposomal Annamycin in Children and Young Adults With Refractory or Relapsed Acute Lymphocytic Leukemia and Acute Myelogeneous Leukemia
Brief Title: Liposomal Annamycin in Children and Young Adults With Refractory or Relapsed ALL or AML
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Participants are no longer being examined or treated.
Sponsor: Callisto Pharmaceuticals (Industry)
Responsible Party: Gary Jacob, Callisto Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-105
Record Dates: First submitted 2007-01-30; First posted 2007-02-01 (Estimated); Last update posted 2011-08-31 (Estimated); Status verified 2011-08

CONDITIONS: Acute Lymphocytic Leukemia; Acute Myelogenous Leukemia
Keywords: Acute Lymphocytic Leukemia; Acute Myelogenous Leukemia; Annamycin; Liposomal Annamycin
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Liposomal Annamycin — 3-day IV infusion

SUMMARY:
This is a Phase I, multi-center, open-label, dose escalation, MTD study of liposomal annamycin in children and young adults with refractory or relapsed ALL or AML. Enrollment will occur in cohorts of approximately 3 subjects with 10 additional subjects enrolled at the MTD. The liposomal annamycin doses will be escalated in sequential cohorts. Six dose levels of liposomal annamycin are planned: 130, 160, 190, 230, 280, and 310 mg/m2/day.The primary objectives of this study are 1) to evaluate the safety and identify the maximum tolerated dose (MTD) of liposomal annamycin when given in 3 consecutive daily doses, starting at 130 mg/m2/day and ranging to as high as 310 mg/m2/day, or the MTD, whichever is lower, in children and young adults with refractory or relapsed acute lymphocytic leukemia (ALL) or acute myelogenous leukemia (AML), and 2) to evaluate the antileukemic activity of liposomal annamycin in children and young adults with refractory or relapsed ALL or AML. The secondary objective is to measure the pharmacokinetics of annamycin and its metabolite, annamycinol.

DETAILED DESCRIPTION:
This is a Phase I, multi-center, open-label, dose escalation, MTD study of liposomal annamycin in children and young adults with refractory or relapsed ALL or AML. Enrollment will occur in cohorts of approximately 3 subjects with 10 additional subjects enrolled at the MTD. The liposomal annamycin doses will be escalated in sequential cohorts. Six dose levels of liposomal annamycin are planned: 130, 160, 190, 230, 280, and 310 mg/m2/day.

The initial group of 3 subjects will receive a treatment cycle of 130 mg/m2/day liposomal annamycin daily for 3 consecutive days followed by 18 days off liposomal annamycin (i.e., 1 treatment cycle = 21 days). A prophylactic mouthwash for use with anthracyline-based chemotherapies (composition described below under Test Product, Dose, and Mode of Administration) will be used 4 times a day on Days 1-4, with one of the 4 times being immediately 1 hour prior to liposomal annamycin treatment on Days 1 3, to prevent oral mucositis. Anti-allergic pre-medication with diphenydramine will be administered before each dose of liposomal annamycin.

Provided that no subject experiences dose limiting toxicity (DLT) [defined as a study drug related Grade 3 or higher non-hematologic toxicity using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v3.0] during the first 21 days (i.e., during the first treatment cycle), the subsequent group of 3 subjects will receive the next higher liposomal annamycin dose. However, if 1 of the 3 initial subjects experiences DLT, the cohort of subjects at the initial dose level will be expanded to 6 subjects. If at least 2 of the 6 subjects experience DLT, then 3 subjects will be treated at the next lower dose. The MTD is defined as the highest dose of liposomal annamycin at which fewer than 2 (of a cohort of up to 6) subjects experience a DLT.

Subsequent dose escalation will occur in a similar fashion. If a subject discontinues treatment for reasons other than study drug related adverse events such that safety cannot be fully evaluated, an additional subject may be enrolled; these will be reviewed on a case-by-case basis in conjunction with the Sponsor. The dose will be escalated until either a MTD is identified or the maximum dose, 310 mg/m2/day, is achieved. Ten additional subjects will be enrolled at the MTD to better define toxicity and to better evaluate efficacy at the MTD.

Subjects will be evaluated before the start of liposomal annamycin treatment and during the first 3 days of liposomal annamycin treatment. Subjects will be evaluated weekly thereafter during the first cycle of treatment (1 cycle consists of 3 weeks, with 3 consecutive days of daily liposomal annamycin treatment followed by 18 days off of liposomal annamycin) and weekly during each subsequent cycle that they are eligible to receive further treatment. A follow-up visit will be conducted 1 to 2 weeks after the final treatment cycle or after the last study drug administration, if the treatment period was prematurely terminated.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of refractory or relapsed ALL or AML.
2. 12 months to 21 years of age at the time of informed consent.
3. Weight ≥10 kg
4. No chemotherapy, radiation, or major surgery within 2 weeks prior to first dose of study drug and recovered from the toxic side effects of such therapy. In the instance of rapidly progressive disease, anti-leukemia therapy may be administered within the 2-week period as long as the subject has recovered from the toxic effects of that therapy. Also, intrathecal therapy may be administered within the 2-week period for subjects with CNS disease.
5. No stem cell transplant regimen within 3 months prior to first dose of study drug.
6. No conventional granulocyte colony stimulating factor (G-CSF) within 7 days prior to the first dose of study drug, and no long-acting G-CSF (Neulasta) within 14 days prior to the first dose of study drug.
7. No investigational therapy within 4 weeks prior to first dose of study drug.
8. Karnofsky Performance Status ≥50% for subjects ≥10 years of age and Lansky Performance Status ≥60% for subjects <10 years of age. Subjects who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance status.
9. Adequate liver function [bilirubin ≤2 times the upper limit of normal (ULN) and serum glutamic-pyruvic transaminase (SGPT) ≤5 times the ULN].
10. Adequate renal function (creatinine clearance ≥60 ml/min/1.73m2).
11. Adequate cardiac function [ejection fraction (EF) >50% or shortening fraction (SF) >28% by echocardiogram or MUGA]
12. Informed consent signed by subject or legal guardian per investigational site guidelines.
13. Able to comply with the requirements of the protocol.
14. Females of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to first dose of study drug.
15. All subjects (male and female) of childbearing potential must agree to practice effective contraception during the entire study period, unless documentation of infertility exists. Should a female become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Exclusion Criteria:

1. Concomitant therapy that includes other chemotherapy that is or may be active against ALL or AML, except for prophylaxis and/or treatment of opportunistic or other infection with antibiotics, antifungals and/or antiviral agents. Concurrent radiation therapy and immunosuppressive therapy are not allowed. Concurrent intrathecal therapy per standard of care is allowed for subjects with CNS disease.
2. Any condition which, in the opinion of the Investigator, places the subject at unacceptable risk if he/she were to participate in the study.
3. Clinically relevant serious co-morbid medical conditions including, but not limited to, active infection, recent (≤6 months) myocardial infarction, unstable angina, symptomatic congestive heart failure, uncontrolled hypertension, uncontrolled cardiac arrhythmias, chronic obstructive or chronic restrictive pulmonary disease, and cirrhosis, or psychiatric illness/social situations that would limit compliance with study requirements. Cardiac patients with a New York Heart Association (NYHA) classification of 3 or 4 will be excluded.
4. Active graft-versus-host disease (GVHD).
5. Pregnant, lactating, or not using adequate contraception.
6. Known allergy to doxorubicin or anthracyclines.
7. Any evidence of mucositis/stomatitis, except for Grade 1 mucositis/stomatitis due to chronic GVHD.

Ages: 12 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2007-02; Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and identify the MTD of liposomal annamycin and to evaluate the antileukemic activity of liposomal annamycin in children and young adults. | 8 months

SECONDARY OUTCOMES:
To measure the pharmacokinetics of annamycin and its metabolite, annamycinol. | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Gary Jacob, Ph.D., Study Director — Callisto Pharmaceuticals, Inc.
Locations (3):
- United States (3):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Denver Children's Hospital, Denver, Colorado
  - Vanderbilt Children's Hospital, Nashville, Tennessee